CLINICAL TRIAL: NCT05178056
Title: Epidural Spinal Cord Stimulation and Respiratory Motor Function After Injury
Brief Title: Spinal Cord Stimulation and Respiration After Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alexander V Ovechkin, MD, PhD, Associate Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21.0564/17.1024; R01HL150581 (NIH)
Record Dates: First submitted 2021-12-01; First posted 2022-01-05 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries; Spinal Cord Stimulation; Breathing Exercises; Rehabilitation
Keywords: Epidural Spinal Cord Stimulation; Respiratory Training
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Our goal is to evaluate the effects of the individually optimized spinal cord Epidural Stimulation (scES) (Aim 1) and to define the efficacy of scES combined with Respiratory Training (RT) (Aim 2) in individuals with Spinal Cord Injury (SCI). Thirty participants with SCI will be recruited, twenty of them will have scES implanted. After screening and recruitment, primary and secondary outcome measurements will be obtained in the Lab at the following time points: 1) Pre intervention, after 30-days without any stimulation and/or intervention, 2) Post mapping, (participants with scES, n=20), 3) Post Session #40 (after 8 weeks of intervention) and 4) Post Session #80 (after 16 weeks of intervention), and 5) Post 16-weeks Follow-up Period. In total, it is anticipated that 5 measurements will be obtained for each participant with implanted scES and 4 measurements for participants without scES.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Respiratory Training (Active Comparator): Research subjects with no implanted stimulator undergoing RT intervention.
  Interventions: Other: Respiratory Training
- Spinal Cord Stimulation (Active Comparator): Research subjects with implanted stimulator undergoing stimulation intervention.
  Interventions: Device: Spinal Cord Epidural Stimulation
- Spinal Cord Stimulation and Respiratory Training (Experimental): Research subjects with implanted stimulator undergoing stimulation intervention in combination with respiratory training.
  Interventions: Device: Spinal Cord Epidural Stimulation; Other: Respiratory Training

INTERVENTIONS:
Device: Spinal Cord Epidural Stimulation — Spinal Cord Epidural Stimulation (scES) will be administered by a multi-electrode array (5-6-5 SpecifyTM electrode, MEDTRONIC, Minneapolis, MN, USA) previously implanted in the epidural space over the dorsum of the spinal cord.
  Arms: Spinal Cord Stimulation; Spinal Cord Stimulation and Respiratory Training
Other: Respiratory Training — Standard threshold Positive Expiratory Pressure Device and standard threshold Inspiratory Muscle Trainer (Respironics Inc., Cedar Grove, NJ) assembled together will be used for respiratory training sessions to complete eighty 45-minute sessions during 16 weeks. The participants will be instructed to perform inspiratory and expiratory efforts against a pressure treshold load.
  Arms: Respiratory Training; Spinal Cord Stimulation and Respiratory Training

SUMMARY:
Respiratory motor control deficit is the leading cause of morbidity and mortality in patients with spinal cord injury. The long-term goal of this NIH-funded study is to develop a rehabilitation strategy for respiration in patients with spinal cord injury as a standard of care. Respiratory function in patients with chronic spinal cord injury can be improved by using inspiratory-expiratory pressure threshold respiratory training protocol. However, the effectiveness of this intervention is limited by the levels of functional capacity preserved below the neurological level of injury. Preliminary data obtained for this study demonstrate that electrical spinal cord stimulation applied epidurally at the lumbar level in combination with respiratory training can activate and re-organize spinal motor networks for respiration. This study is designed to investigate respiratory motor control-related responses to epidural spinal cord stimulation alone and in combination with respiratory training. By characterization of respiratory muscle activation patterns using surface electromyography in association with pulmonary functional and respiration-related cardiovascular measures, the investigators expect to determine the specific stimulation parameters needed to increase spinal excitability below level of injury to enhance responses to the input from supraspinal centers that remain after injury and to promote the neural plasticity driven by the respiratory training. This hypothesis will be tested by pursuing two Specific Aims: 1) Evaluate the acute effects of epidural spinal cord stimulation on respiratory functional and motor control properties; and 2) Evaluate the effectiveness of epidural spinal cord stimulation combined with respiratory training.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is commonly associated with motor control deficits. When injury alters the control of trunk muscles, respiratory function is compromised leading to respiratory complications (including COVID19-related), one of the primary causes of morbidity and mortality in patients with chronic SCI. However, none of the respiratory rehabilitative modalities for this population have yet been proven to be clinically effective.

Previous work demonstrated that respiratory motor function can be improved by using inspiratory-expiratory pressure threshold respiratory training protocol. It have been found that these improvements are associated with respiratory motor and autonomic activity-based plasticity. However, due to low excitability of spinal networks below the injury, the effectiveness of this intervention is limited to the levels of functional capacity preserved after injury.

Epidural Stimulation (scES) can activate spinal networks below level of the spinal cord lesion. It was demonstrated that tonic scES at the lumbar level in individuals with SCI lead to voltage-dependent changes in breathing pattern and enhanced voluntary respiratory muscle activation below the injury level. Preliminary data collected for this proposal indicate that spinal cord stimulation can enhance the adaptive plasticity and provide amplified therapeutic effects when it is combined with respiratory training.

The objective of this study is to investigate the mechanisms of respiratory functional and respiratory motor responses to the scES as an important step toward the long-term goal of developing effective evidence-based rehabilitation strategies for patients with SCI. The central hypothesis is that scES raises the excitability of motor networks for respiration resulting in amplified use-dependent neural plasticity in response to the respiratory training. The rationale for the proposed study is to justify the development of a new direction in respiratory rehabilitation by using respiratory training in combination with electrical spinal cord stimulation.

The central hypothesis will be tested by pursuing the following two specific aims:

Specific Aim 1: Evaluate the acute effects of epidural spinal cord stimulation on respiratory functional and motor control properties.

Hypothesize is that the scES increases spinal motor network excitability leading to increased respiratory functional outcomes due to enhanced activation of neural networks specific for respiration. A comparative approach focusing on clinical and electrophysiological characterizations of respiratory functional and motor control responses in the presence or absence of scES in individuals with high-level chronic SCI will be used. Respiratory motor control will be characterized by using pulmonary function test, electromyography and recordings of trunk kinematics assessed during respiratory efforts. During these assessments, beat-to-beat blood pressure and heart rate / respiratory rate variability will be assessed to evaluate respiratory-cardiovascular interactions.

Specific Aim 2: Evaluate the effectiveness of epidural spinal cord stimulation combined with respiratory training.

Hypothesis is that specifically configured scES combined with respiratory training allows enhanced use-dependent neural plasticity for respiration. This hypotheses will be confirmed if the respiratory training combined with scES results in significantly improved functional outcomes when compared to the measures obtained from either scES-only or respiratory training-only groups. The physiological characterization of respiratory functional and motor control responses in these groups will be used to identify specific therapeutic effects. This work will be done by using methods outlined in Aim 1 and additional clinical measures all assessed before/after stimulation and/or training and during the follow-up period.

This randomized, controlled clinical trial will evaluate the effects of the scES approach to target respiratory neural networks and will test the rehabilitative capacity of respiratory activity-based training in combination with spinal cord stimulation applied epidurally. Such results are expected to have an important positive impact, because, for the first time, identified effects of this strategy will provide evidence that respiratory function can be effectively restored in patients with severe chronic SCI.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Stable medical condition
* Non-progressive C3-T1 AIS A-C Spinal Cord Injury (SCI)
* Sustained SCI at least 24 months prior to entering the study
* At least 15%-deficit in pulmonary function outcomes

Exclusion Criteria:

* Painful musculo-skeletal dysfunction
* Unhealed fracture
* Contracture
* Pressure sore
* Urinary tract infection that might interfere with respiratory training
* Clinically significant depression
* Psychiatric disorders
* Ongoing drug abuse;
* Major cardiovascular disease
* Major pulmonary disease
* Ventilator dependence
* Major endocrine disorders
* Malignancy
* Marked obesity
* Deep vein thrombosis
* HIV/AIDS related illness
* Secondary causes of respiratory dysfunction
* Major gastrointestinal problems
* Other major medical illness contraindicated for respiratory training
* Pregnantcy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Maximum Expiratory Pressure (PEmax) | Through study completion, an average of 1 year.
  Standard Spirometry measurement.
Change in Surface electromyography (sEMG) Magnitude (Mag) | Through study completion, an average of 1 year.
  Respiratory multi-muscle activation measures assessed using standard surface electromyography.
Change in Surface electromyography (sEMG) Similarity Index (SI) | Through study completion, an average of 1 year.
  Respiratory multi-muscle activation measures assessed using standard surface electromyography.
Change in Maximum Inspiratory Pressure (PImax) | Through study completion, an average of 1 year.
  Standard Spirometry measurement.

SECONDARY OUTCOMES:
Change in Forced Vital Capacity (FVC) | Through study completion, an average of 1 year.
  Standard Spirometry measurement.
Change in Forced Expiratory Volume in 1 second (FEV1) | Through study completion, an average of 1 year.
  Standard Spirometry measurement.
Change in Baroreflex sensitivity (BRS) | Through study completion, an average of 1 year.
  Measure of the beat-to-beat blood pressure and heart rate variability assessed during a Valsalva maneuver and maximum respiratory effort.
Change in Baroreflex Effectiveness Index (BEI) | Through study completion, an average of 1 year.
  Measure of the beat-to-beat blood pressure and heart rate variability assessed during a Valsalva maneuver and maximum respiratory effort.

OTHER OUTCOMES:
Changes in Spinal Cord Independence Measure (SCIM) scores | Through study completion, an average of 1 year.
  The SCIM (version III) measures the levels of self-care and mobility.
Changes in The Craig Handicap Assessment & Reporting Technique (CHART) scores | Through study completion, an average of 1 year.
  The CHART measure the level of handicap in a community setting: physical independence, mobility, occupation, social integration, economic self-sufficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ovechkin, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- Frazier Rehabilitation and Neuroscience Institute, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No